CLINICAL TRIAL: NCT01823419
Title: Omega-6 to Omega-3 Fatty Acid Ratio and Higher Order Cognitive Function in 7-to 9-year-olds
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Carol Cheatham, PhD, Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: 10-1401
Record Dates: First submitted 2013-03-20; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Typical Development

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 7-9 year olds: Typically developing 7- to 9-year-olds will be enrolled and tested.

SUMMARY:
The purpose of this study is to investigate the role of the ratio of omega-6 to omega-3 fatty acids on executive functions. The investigators hypothesize that participants ages 7-9 years with a ratio closer to 4:1 will do better on tests of executive function than participants with a ratio closer to the purported Western diet norm of 15:1.

ELIGIBILITY:
Inclusion Criteria:

* typically-developing

Exclusion Criteria:

* not fluent in English

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 7-9 year olds
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Relation between executive function and n-6/n-3 fatty acid intake | up to 10 days
  Executive function will be measured using a validated and standardized system known as CANTAB (Cambridge Neuropsychological Test Automated Battery) and correlated with the ratio of fatty acid intake. 24-hour diet recalls will be completed using the NDSR (Nutrient Data System for Research) software. Across one week, the children will be interviewed 3 times (two weekdays, one weekend day) about what they ate in the previous 24 hours. The dietary data will be averaged to arrive at the n-6/n-3 intake. The children will then come to lab for one visit where they will be assessed using the CANTAB.

SECONDARY OUTCOMES:
Temperament | Baseline
  Temperament will be measured using a Rothbart written assessment completed by the caregiver.
Socioeconomic status | Baseline
  Demographic information will be collected from caregiver using a lab-typical questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Cheatham, PhD, Principal Investigator — UNC-Chapel Hill; Kelly W Sheppard, BS, Study Director — UNC-Chapel Hill
Locations (1):
- UNC at Chapel Hill Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Sheppard KW, Cheatham CL. Omega-6/omega-3 fatty acid intake of children and older adults in the U.S.: dietary intake in comparison to current dietary recommendations and the Healthy Eating Index. Lipids Health Dis. 2018 Mar 9;17(1):43. doi: 10.1186/s12944-018-0693-9. PMID 29523147
- [Derived] Sheppard KW, Cheatham CL. Omega-6 to omega-3 fatty acid ratio and higher-order cognitive functions in 7- to 9-y-olds: a cross-sectional study. Am J Clin Nutr. 2013 Sep;98(3):659-67. doi: 10.3945/ajcn.113.058719. Epub 2013 Jul 3. PMID 23824723